CLINICAL TRIAL: NCT07240207
Title: Dissecting Tumour MicroenvirOnment in Solid Paediatric Tumour to Improve Adoptive Cell Therapy
Acronym: MOST
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Mirko Bertozzi, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: MOST
Record Dates: First submitted 2025-09-11; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Solid Tumors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Pediatric solid tumors exhibit a low mutational burden, limited availability of neoantigens, and poor infiltration of tumor-infiltrating lymphocytes (TILs) within the tumor microenvironment (TME), characteristics that reduce the effectiveness of immunotherapies in children. However, pediatric tumors express a subgroup of antigens that can be exploited as targets. Stimulating the T lymphocyte response against these antigens could overcome immunosuppressive barriers. The adoption of therapies based on cytotoxic T lymphocytes (CTLs) represents a promising strategy.

A total of 42 neoplasms were analyzed, including: 8 neuroblastomas, 7 sarcomas, 4 nephroblastomas, 1 renal carcinoma, 2 rhabdomyosarcomas, 5 lymphomas, 2 ovarian carcinomas, 4 teratomas, 2 thyroid tumors, and 7 other rare tumors. Primary cells from these tumors were preserved, resulting in the stabilization of 5 cell lines used for functional studies in vitro.

Currently, 4 tumor-specific CTL lines derived from healthy adult donors have been expanded; tumor antigen-specific T cells showed the ability to recognize and kill commercial tumor cell lines as well as stabilized pediatric tumor lines from osteosarcoma, nephroblastoma, and neuroblastoma. In particular, the G-Rex bioreactor enabled greater expansion of CTLs while maintaining a broad spectrum of specificity for most tumor antigens and a lymphocyte phenotype with an increased composition of early memory T cells, correlated with greater persistence in vivo.

The results demonstrate that the use of bioreactors represents a significant advancement in the production of CTLs specific for pediatric tumor antigens. The ability of CTLs derived from bioreactors to express early memory and activation markers makes them particularly promising for clinical applications, where persistence and efficacy are key factors.

Based on the presented results, the analysis of in vivo persistence and cytotoxic capacities in preclinical models will be deepened, aiming to confirm the efficacy of the produced cells.

The main objective of the project is to develop expansion protocols for CTLs specific to pediatric tumor antigens, proposing innovative protocols for the ex vivo expansion of CTLs targeting pediatric tumor antigens.

Finally, standardizing the large-scale process could be another necessary objective to translate these findings into practical clinical applications improving immunotherapy in pediatric cancer with evident benefits for affected children and care givers.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients 0-18 years
* affected by solid tumors

Exclusion Criteria:

* patients over 18
* non-solid malignancies

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients affected by solid tumors enrolled for treatment at Fondazione IRCCS Policlinico San Matteo, pavia, Italy in the period 2023-2025
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cytotoxic Activity of Expanded CTLs Against Pediatric Tumor Cell Lines In Vitro | Days 7, 14, and 21 post-CTL expansion
  Cytotoxic activity of tumor antigen-specific cytotoxic T lymphocytes (CTLs) expanded using G-Rex bioreactors will be measured by quantifying target cell lysis using a standard chromium-51 release assay or flow cytometry-based killing assay against stabilized pediatric tumor cell lines, including neuroblastoma, nephroblastoma, and osteosarcoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Chirurgia Pediatrica, Pavia, Pavia, Italy